CLINICAL TRIAL: NCT04697446
Title: An External Control, Observational, Retrospective Study Assessing the Effect of Pralsetinib Compared With Best Available Therapy for Patients With RET-Fusion Positive Advanced Non-Small Cell Lung Cancer
Brief Title: External Control, Observational, Retrospective Study Comparing Pralsetinib to Best Available Therapy in Patients With RET-Fusion Positive NSCLC
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Blueprint Medicines Corporation (Industry)
Collaborators: Analysis Group, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BLU-667-2404
Record Dates: First submitted 2020-12-16; First posted 2021-01-06 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: RET-fusion Non Small Cell Lung Cancer; Lung Neoplasm; Carcinoma, Non-Small-Cell Lung; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Lung Diseases; Respiratory Tract Diseases; Carcinoma, Bronchogenic; Bronchial Diseases; Head and Neck Neoplasms; Carcinoma; Neoplasms by Histologic Type; Neoplasms, Germ Cell and Embryonal; Neoplasms, Nerve Tissue; Metastatic Non Small Cell Lung Cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Lung Diseases; Respiratory Tract Diseases; Carcinoma, Bronchogenic; Bronchial Diseases; Head and Neck Neoplasms; Carcinoma; Neoplasms by Histologic Type; Neoplasms, Germ Cell and Embryonal; Neoplasms, Nerve Tissue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients from the BLU-667-1101 (ARROW) study: Patients with Non-Small Cell Lung Cancer (NSCLC) who received treatment with pralsetinib as part of the BLU-667-1101 (ARROW) study
- External Control Group: Patients with Non-Small Cell Lung Cancer (NSCLC) that received best available therapy

SUMMARY:
This is an external control, observational, retrospective study designed to compare clinical outcomes for pralsetinib compared with best available therapy for patients with RET-fusion positive advanced NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Must have a diagnosis of locally advanced (non-resectable) or metastatic RET-fusion positive NSCLC
* Must have received at least one line of systemic therapy for locally advanced (non-resectable) or metastatic RET-fusion positive NSCLC, which may include regimens containing:

  * Chemotherapy, e.g., regimens containing platinum doublet-based therapy (carboplatin, cisplatin)
  * Chemotherapy in combination with other drugs will be assessed, e.g., in combination with pemetrexed, immune checkpoint inhibitors (pembrolizumab), bevacizumab
  * Ramucirumab in combination with docetaxel
  * Immune checkpoint inhibitors, e.g., pembrolizumab, nivolumab, and atezolizumab
  * MKIs, e.g., cabozantinib, alectinib, vandetanib, sunitinib, and nintedanib
* Must be aged ≥18 years of age at the initiation of first systemic line of therapy
* Must have availabile of performance status (e.g., Eastern Cooperative Oncology Group [ECOG] score or Karnofsky score)
* Must have an index date at least 3 months prior to the start of data collection (in order to include patients with at least 3 months of follow-up after index date), unless date of death occurred less than three months from index date
* Must have an approved waiver of informed consent or signed informed consent for participation in the retrospective chart review study, as applicable

Exclusion Criteria:

* Known primary driver alteration other than RET (e.g., targetable mutation in EGFR, ALK, ROS1, or BRAF)
* History of other malignancy, other than non-melanoma skin cancer, within 1 year prior to initiation of first systemic therapy
* Received pralsetinib as the first line of systemic therapy for RET-fusion positive NSCLC, or prior to initiation of first systemic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include patients with locally advanced or metastatic RET-fusion positive non-small cell lung cancer (NSCLC)
Sampling Method: Probability Sample
Enrollment: 279 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Comparative evaluation of real-world response rate (rwORR) between patients receiving best available therapy versus pralsetinib | Up to 12 years
  rwORR, defined as the proportion of patients with clinician-assess complete response (CR) or partial response (PR)

SECONDARY OUTCOMES:
Comparative evaluation between patients receiving best available therapy versus pralsetinib of Overall survival (OS) | Up to 12 years
  OS, defined as time from initiation of a given line of therapy to death from any cause
Comparative evaluation between patients receiving best available therapy versus pralsetinib of Real-world duration of response (rwDOR) | Up to 12 years
  rwDOR, defined as the duration of time from the first documented clinician-assessed response to the first documented clinician-assessed progressive disease or death due to any cause within 30 days of the last radiological exam, for each line of treatment
Comparative evaluation between patients receiving best available therapy versus pralsetinib of Real-world disease control rate (rwDCR) | Up to 12 years
  rwDCR, defined as proportion of patients with clinician-assessed complete response, partial response, or stable disease
Comparative evaluation between patients receiving best available therapy versus pralsetinib of Real-world clinical benefit rate (rwCBR) | Up to 12 years
  rwCBR, defined as proportion of patients who had documented clinician-assessed complete response or partial response, or stable disease lasting at least 16 weeks
Comparative evaluation between patients receiving best available therapy versus pralsetinib of Real-world progression-free survival (rwPFS) | Up to 12 years
  rwPFS, defined as time from initiation of line of therapy to clinician-assessed disease progression or death from any cause, whichever occurs first
Comparative evaluation between patients receiving best available therapy versus pralsetinib of Duration of treatment (DOT) | Up to 12 years
  DOT, defined as time from initiation of line of systemic treatment to discontinuation of same line of treatment for any reason
Comparative evaluation between patients receiving best available therapy versus pralsetinib of Time to next treatment line (TtNTL) | Up to 12 years
  TtNTL, defined as the time from initiation of line of systemic treatment to the initiation of the next line of treatment
To characterize the safety profile and conduct comparative evaluation of safety between patients receiving best available care vs. pralsetinib | Up to 12 years
  Adverse events (AEs) that result in treatment modification or discontinuation, hospitalization, or death according to evaluation of responsible physician

CONTACTS AND LOCATIONS:
Locations (3):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States
- University Hospital Center of Toulouse - Larrey Hospital, Toulouse, France
- Lucerne Cantonal Hospital, Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No